CLINICAL TRIAL: NCT06785363
Title: Effect of Pumped Technique for Ilio-lumber Ligament Release on Postnatal Low Back Pain
Brief Title: The Study Focuses on the Release of the Iliolumbar Ligament Using a Pumped Technique, Addressing Its Tightness Caused by Excessive Anterior Pelvic Tilt During Pregnancy. This Condition Often Results in Low Back Pain and Mechanical Dysfunction of the Lumbar and Sacroiliac Regions.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moataz Abdelaal Mohamed, Teacher assistance in Faculty of physical therapy, Pharos University in Alexandria, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.Rec/012/005571
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain
Keywords: low back pain; lumbar and sacroiliac pain; iliolumbar ligament disorder
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pumped technique for iliolumbar ligament release (Experimental)
  Interventions: Other: pumped technique for ilio-lumbar ligament release
- Hot packs (Active Comparator): postnatal women will be treated by hot packs for 20 minutes three times per week for 8 weeks.
  Interventions: Other: Hot Packs

INTERVENTIONS:
Other: pumped technique for ilio-lumbar ligament release — Patient position: the patient lying supine or side lying Therapist position: standing on one side of patient. Hand grip: one hand placed on posterior region of iliac crest (close to attachment of ilio-lumbar ligament) while other hand stabilize the medial part of thigh. Therapist force: therapist pulling patient's thigh posteriorly.
  Arms: Pumped technique for iliolumbar ligament release
Other: Hot Packs — postnatal women will be treated by hot packs for 20 minutes three times per week for 8 weeks.
  Arms: Hot packs

SUMMARY:
The iliolumbar ligament, one of the sacroiliac ligaments, has been identified in recent research as a contributor to low back pain when tight. During pregnancy, hormonal changes and postural changes can cause this ligament to tighten, leading to pain. Releasing the iliolumbar ligament can reduce low back pain and restore normal mechanical function.

DETAILED DESCRIPTION:
Group A (Control group) It will be consisted of postnatal women and will be treated by hot packs for 20 minutes three times per week for 8 weeks.

Group B (study group) the participant will treated by hot packs for 20 min in additional to pumping technique for iliolumbar ligament release for 30 min. 3 times per week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1- the women are delivery within 3 months. 3- Their BMI must be less than 30 Kg\m 2 . 4- Its included primipara or multipara. 5- Its included be normal vaginal labor delivery or caesarian section.

Exclusion Criteria:

1. Clinical diagnosis by Lumbar disc prolapse.
2. Clinical diagnosis by Lumbar spondylolysis and spondlysis.
3. Clinical diagnosis by back trauma or fracture.
4. Clinical diagnosis by Lumbar canal stenosis.
5. Clinical diagnosis by Rheumatoid arthritis.
6. Clinical diagnosis by Malignancy.
7. Clinical diagnosis by any deformity for low limb.
8. Clinical diagnosis by Scoliosis.
9. Taking analgesic drugs.
10. Clinical diagnosis by Deep vein thrombosis

Ages: 25 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS): | 8 weeks
  It will be used to assess the severity of low back pain in women from both groups A and B before and after treatment. The scoring ranges from 1, indicating the least pain and discomfort, to 10, representing the most severe pain and discomfort.
Goniometer | 8 weeks
  It will be used to assess lumbar flexion range of motion for each woman in both groups A and B before and after treatment.
Inclinometer | 8 weeks
  It will be used to assess lumbar curvature for each woman in both groups A and B before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://mtprehabjournal.emnuvens.com.br/revista/article/view/769